CLINICAL TRIAL: NCT03735316
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study for High-Dose Hydroxocobalamin (Vitamin B12A) for Vasopressor Refractory Hypotension Following Cardiopulmonary Bypass
Brief Title: Vitamin B12a Vasoplegic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment over study period
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James A. Nelson, Principle Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17-011130
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Vasoplegic Syndrome
Keywords: Vitamin B12a; Hypotension; Cardiopulmonary Bypass
MeSH Terms: conditions — Vasoplegia; Hypotension | interventions — Hydroxocobalamin; Vitamin B 12; Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking and blinding will be carried out by the research pharmacy with unmasking to be performed at study completion through the research pharmacy and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- B12a (Experimental): Subjects will receive Hydroxocobalamin marketed as Cyanokit®, 5g, IV
  Interventions: Drug: Hydroxocobalamin; Procedure: Cardiopulmonary Bypass
- Placebo (Placebo Comparator): Subjects will receive placebo
  Interventions: Procedure: Cardiopulmonary Bypass; Drug: Placebos

INTERVENTIONS:
Drug: Hydroxocobalamin — 5g, IV, Infused once over 15 minutes. The drug comes in a 250ml glass vial with 5g of lyophilized hydroxocobalamin to be reconstituted in 200ml of Normal Saline, Dextrose or Lactated Ringers.
  Other Names: Cyanokit®, Vitamin B12a
  Arms: B12a
Procedure: Cardiopulmonary Bypass — Technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the patient's body.
  Other Names: CPB
Drug: Placebos — Placebo is a Normal Saline, 5g, IV, Infused once over 15 minutes. The placebo comes in a 250ml glass vial.
  Arms: Placebo

SUMMARY:
The study team will evaluate the medication Hydroxocobalamin (B12a) for treatment of low blood pressure after cardiac surgery.

DETAILED DESCRIPTION:
If subjects meet the criteria for inclusion in the study based on the subjects blood pressure the subject will be randomized to receive the study drug or a placebo. Subjects blood pressure will be monitored closely for the first 30 minutes and then have standard intensive care unit (ICU) care afterwards. Kidney dysfunction will be assessed for changes in urine production and laboratory values that are followed as a part of standard postoperative care. Study coordinators will obtain these values from subjects medical records for 7 days and subjects will be contacted by phone for follow up after 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Any patient for whom we are able to obtain consent ahead of their procedure
* Patients presenting for a procedure in which cardiopulmonary bypass will be required
* Considered high risk for vasoplegic syndrome
* Has no contraindications to arterial line or PA catheter placement
* Develops high-dose vasopressors for 30 min or longer and refractory hypotension consistent with vasoplegic syndrome within 24 hours of coming off cardiopulmonary bypass.

Exclusion Criteria:

* Age<18 years
* Known pregnancy or patients without a documented pregnancy test if not menopausal.
* Known prior anaphylactic or allergic reaction to B12a
* CKD stage 4 or worse
* ECMO (extracorporeal membrane oxygenation) prior to study consent.
* Patients currently on cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Nelson, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Saint Mary's Hospital, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- B12a: Subjects received Hydroxocobalamin marketed as Cyanokit®, 5g, IV
  Hydroxocobalamin: 5g, IV, Infused once over 15 minutes. The drug comes in a 250ml glass vial with 5g of lyophilized hydroxocobalamin to be reconstituted in 200ml of Normal Saline, Dextrose or Lactated Ringers.
  Cardiopulmonary Bypass: Technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the patient's body.
- Placebo: Subjects received placebo
  Cardiopulmonary Bypass: Technique that temporarily takes over the function of the heart and lungs during surgery, maintaining the circulation of blood and the oxygen content of the patient's body.
  Placebos: Placebo is a Normal Saline, 5g, IV, Infused once over 15 minutes. The placebo comes in a 250ml glass vial.
Period: Overall Study
Arm/Group | B12a | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B12a | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [56 to 69] | 70 [64 to 73] | 69 [60 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Pressure
Description: The average pressure in a patient's arteries during one cardiac cycle
Time Frame: baseline, 4 hours
Population: Terminated study. Insufficient recruitment over study period
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
mmHg | 6 [1.25 to 9.5] | -0.5 [-2.75 to 1.25]

2. Secondary Outcome: Change in Norepinephrine Equivalent Infusion Rate. Norepinephrine Equivalent Table is Listed in the Study Protocol
Description: Vasopressors are administered and adjusted to maintain blood pressure. The combined dose of vasopressor dosage was calculated as norepinepheine equivalents listed in Table 1 of the protocol appendix and measured as a secondary outcome through the first 4 hours after intevention.
Time Frame: baseline, 4 hours
Population: Terminated study. Insufficient recruitment over study period
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
mcg/kg/min | -0.035 [-0.0625 to -0.0150] | 0.02 [0.0075 to 0.0425]

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: The maximum arterial pressure during contraction of the left ventricle of the heart.
Time Frame: baseline, 4 hours
Population: Terminated study. Insufficient recruitment over study period
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
mmHg | 5.5 [-0.5 to 9.75] | 0.5 [-1.25 to 1.25]

4. Secondary Outcome: Death
Description: Number subject deaths
Time Frame: 30 days
Population: Terminated study. Insufficient recruitment over study period
Measure: Count of Participants; unit: Participants
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

5. Secondary Outcome: Duration of Hospital Stay
Description: Number of days subjects are hospitalized
Time Frame: 30 days
Population: Terminated study. Insufficient recruitment over study period
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
days | 11.5 [8 to 16.5] | 15 [12.5 to 18.0]

6. Secondary Outcome: Duration of Intensive Care Stay
Description: Number of days subjects are in the intensive care unit
Time Frame: 30 days
Population: Terminated study. Insufficient recruitment over study period
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | B12a | Placebo
Number analyzed (Participants) | 4 | 4
days | 6 [3.75 to 9.5] | 8.50 [6.5 to 9.25]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 30 days
Arm/Group | B12a | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B12a (N=4) | Placebo (N=4)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Terminated study. Insufficient recruitment over study period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03735316/Prot_SAP_000.pdf